CLINICAL TRIAL: NCT05252156
Title: An Open-label Randomized Controlled Trial Assessing the Efficacy of Two Levels of Intraoral Neuromuscular Electrical Stimulation for Moderate Obstructive Sleep Apnea: The ELMO Trial
Brief Title: eXciteOSA for Treatment of Moderate Obstructive Sleep Apnea
Acronym: ELMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Signifier Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMT_EOSA_SZT_0003
Record Dates: First submitted 2022-02-12; First posted 2022-02-23 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Therapy Dose-A (Experimental): Neuromuscular electrical stimulation; two 20-minute sessions per day.
  Interventions: Device: eXciteOSA
- Therapy Dose-B (Experimental): Neuromuscular electrical stimulation; one 30-minute session per day.
  Interventions: Device: eXciteOSA
- No Therapy (No Intervention): Under the care of the referring physician, with no therapy applied

INTERVENTIONS:
Device: eXciteOSA — eXciteOSA
  Arms: Therapy Dose-A; Therapy Dose-B

SUMMARY:
The objective of this study is to assess the efficacy of the eXciteOSA device amongst a sample of patients with moderate OSA. The study is a multi-center, prospective, open-label, randomized, parallel-arm trial of eXciteOSA (administered at two doses) versus no-therapy for six weeks. Up to 120 participants will be enrolled, in order to randomized n=62.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=18 years;
* Diagnosed with moderate OSA;
* Smartphone or tablet capable of running the eXciteOSA app;
* Fluent in written and spoken English.

Exclusion Criteria:

* BMI >=35 kg/m2;
* Implanted medical device;
* Dental braces and/or intraoral metal jewelry;
* Any condition impacting the tissue of the oral cavity, including but not limited to ulceration or periodontitis;
* Symptomatic nasal pathology such as septal deviation, nasal polyposis, or chronic rhinosinusitis;
* Tonsillar hypertrophy (tonsil size grade 3 or greater);
* Clinically significant facial or oropharyngeal abnormalities such as class 2 malocclusion;
* Prior oropharyngeal surgery for sleep-disordered breathing;
* At-home use of a mandibular advancement device or PAP for sleep-disordered breathing within the previous four weeks;
* Use of any overnight therapy that cannot be withdrawn during study enrollment;
* Diagnosed with any sleep disorder other than OSA;
* Chronic use of central nervous system depressants;
* Driver in a sleepiness-related vehicular accident or near-miss within the two years prior to enrolment (self-report);
* Employed as a commercial driver, pilot, or other occupation that may be impacted by hypersomnolence;
* Considered by the PI to be at risk of an AE resulting from hypersomnolence;
* Any periods of non-connectivity (wifi or cellular data) exceeding 48 hours planned to take place, or likely to take place, during enrollment;
* Current or planned pregnancy;
* Member of a vulnerable population, including but not limited to prisoners and those lacking consent capacity;
* Clinically-significant burden of comorbidities (including history of myocardial infarction, cardiac arrhythmia, heart failure, history of stroke, or transient ischemic attack), and/or any other limitation or condition that may impact the patient's ability to complete the study protocol and use the device per the Instructions for Use (PI discretion);
* Employee and/or residing household member who is an employee of a company that produces or distributes products designed to diagnose, treat, and/or monitor sleep or sleep-disordered breathing (including the Sponsor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The difference in the delta-REI (baseline to follow-up) between therapy (Dose-A and Dose-B combined) and no therapy | Six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Zayni, Study Director — yasser.z@signifiermedical.com
Locations (7):
- United States (7):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Delta Waves, Colorado Springs, Colorado
  - Florida Lung & Sleep Associates, Lehigh Acres, Florida
  - Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland
  - Clayton Sleep Institute, St Louis, Missouri
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Bogan Sleep Consultants, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No